CLINICAL TRIAL: NCT06109363
Title: Effectiveness of a Stepped Care Model to Deliver Cognitive-behaviour Therapy for Insomnia in Adults, a Pragmatic Stepped-wedge Cluster Randomized Trial
Brief Title: A Stepped Care Model to Deliver CBT-I in Community
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Wing Yun Kwok, Professor, Department of Psychiatry, Chinese University of Hong Kong
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 20230816
Record Dates: First submitted 2023-10-13; First posted 2023-10-31 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Insomnia; Sleep Disturbance
Keywords: Insomnia; Stepped care model; Stepped wedge cluster randomized trial
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Parasomnias | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Pragmatic stepped wedge design - over 4 months, 18 sites enter trial at 1 month intervals. 2
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Stepped-care CBT-I group (Experimental): A total of 3 steps of CBT-I intervention will be provided, with the objectives to increase the awareness of sleep health, increase sleep literacy, establish good sleep hygiene and treat insomnia.
  Step 1: self-help digital CBT-I program; Step 2: guided CBT-I program; Step 3: individualized consultation.
  Interventions: Behavioral: Cognitive behavioral therapy for insomnia (CBT-I)
- Control group (No Intervention): Participants in the control group remain unexposed to the stepped-care CBT-I intervention.

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy for insomnia (CBT-I) — CBT-I intervention will be provided to participants once their districts are exposed.
  Arms: Stepped-care CBT-I group

SUMMARY:
Insomnia is one of the most common sleep disorders and affects approximately 10 - 40% of the population across different age groups in Hong Kong. Cognitive behavioral therapy for insomnia (CBT-I) is the first line treatment for adult insomnia due to its comparable effect to medication in short term but is more sustainable in the long run. However, only a few sufferers have received CBT-I, due to limited accessibility, lack of trained sleep therapists, time costing and geographical limitations. To increase CBT-I accessibility, different formats of CBT-I have been proposed. Empirical evidence including ours consistently suggested that self-help digital CBT-I is effective in improving sleep while its augmentation with a guided approach could further enhance the treatment gain. Previous evidence has suggested that although self-help CBT-I could lead to positive outcomes, the drop out rate is quite high and maybe less effective for patients with comorbidity or high level of distress.

Thus, a stepped-care approach to CBT-I that utilizes online self help and therapist-guided modes of delivery might be a potential way to facilitate efficient dissemination of effective insomnia treatment resources. The effectiveness of the stepped care model will be evaluated in a real world setting using stepped-wedge cluster randomized controlled design. The program will be rolled out to different districts in Hong Kong sequentially in 18 districts over 4 steps with a eqaully spaced time periods.

DETAILED DESCRIPTION:
This interventional study will be a multicenter, assessor-blinded, pragmatic stepped-wedge cluster randomized controlled trial. A total of 18 districts will be included in the study and the randomization will be carried out based on the districts. The stepped-care CBT-I intervention will be sequentially rolled out to the 4-6 districts per step according to a computer-generated random number while the remaining clusters will continue to stay unexposed to the CBT-I intervention over the control period. Therefore after 4-step exposure, all clusters will receive the stepped-care CBT-I intervention. A total of 3 follow-up assessments (post intervention, 3-month and 12-month follow up) will be conducted to assess the effectiveness and long-term effects of the stepped care model.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese adults aged 18-70 years old,
2. The score of Insomnia Severity Index ≥ 10.

Exclusion Criteria:

1. present with psychotic disorders such as bipolar disorder and schizophrenia,
2. present with severe depression or suicidal ideation,
3. present with neurodegenerative diseases that prevent participant from completing the intervention (e.g., dementia and Parkinson's disease).
4. unable to provide consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1100 (Estimated)
Dates: Start 2023-10-23 (Actual); Primary Completion 2026-01-22 (Estimated); Study Completion 2026-04-22 (Estimated)

PRIMARY OUTCOMES:
Insomnia severity index | Post-intervention (ranging from 8 weeks to 24 weeks, depending on the treatment level), 3-month post-intervention and 12-month post-intervention follow up
  The primary outcome will be the perceived insomnia severity measured by Insomnia Severity Index (ISI).

SECONDARY OUTCOMES:
Severity of depression | Post-intervention (ranging from 8 weeks to 24 weeks, depending on the treatment level), 3-month post-intervention and 12-month post-intervention follow up
  Patient Health Questionnaire-9 (PHQ-9) will be used to measure the severity of depression.
Severity of anxiety | Post-intervention (ranging from 8 weeks to 24 weeks, depending on the treatment level), 3-month post-intervention and 12-month post-intervention follow up
  General Anxiety Disorder-7 (GAD-7) will be used to measure the severity of anxiety.
Health-related quality of life | Post-intervention (ranging from 8 weeks to 24 weeks, depending on the treatment level), 3-month post-intervention and 12-month post-intervention follow up
  The health-related quality of life (HRQoL) will be measured by the EuroQol-5D (EQ).
Chronic insomnia diagnosis | Post-intervention (ranging from 8 weeks to 24 weeks, depending on the treatment level), 3-month post-intervention and 12-month post-intervention follow up
  A checklist based on Diagnostic and statistical manual of mental disorders will be implemented to measure the incidence of chronic insomnia.
Medication usage | Post-intervention (ranging from 8 weeks to 24 weeks, depending on the treatment level), 3-month post-intervention and 12-month post-intervention follow up
  A checklist will be used to measure the subject's medication usage change over the past 3 months.
Clinical global impression | Post-intervention (ranging from 8 weeks to 24 weeks, depending on the treatment level), 3-month post-intervention and 12-month post-intervention follow up
  Clinical Global Impression (CGI) will be used to assess the overall improvement or change in a patient's condition over time.
Patient-report clinical global impression | Post-intervention (ranging from 8 weeks to 24 weeks, depending on the treatment level), 3-month post-intervention and 12-month post-intervention follow up
  A single-item CGI will be used to ask the participant whether they experience sleep improvement or change over the past week or not.
Sleep duration | Post-intervention (ranging from 8 weeks to 24 weeks, depending on the treatment level), 3-month post-intervention and 12-month post-intervention follow up
  Two self-report questions will be used to record the sleep duration during weekdays and weekends of the participants.
Subjective sleep as measured by sleep diary | Post-intervention (ranging from 8 weeks to 24 weeks, depending on the treatment level), 3-month post-intervention and 12-month post-intervention follow up
  Self-report sleep diary will be used to record subjective sleep of the participants including total time in bed, sleep onset latency, total sleep duration, sleep efficiency and wake after sleep onset.
Healthcare resource use | Post-intervention (ranging from 8 weeks to 24 weeks, depending on the treatment level), 3-month post-intervention and 12-month post-intervention follow up
  The use and expense of sleep-promoting medication, psychotherapy, and other complementary treatments for sleep improvement over the past 3 months will be collected from individual participants using a self-developed questionnaire, with a focus on their healthcare resource utilization.
Work and social functioning | Post-intervention (ranging from 8 weeks to 24 weeks, depending on the treatment level), 3-month post-intervention and 12-month post-intervention follow up
  A 5-item questionnaire developed from Work and Social Adjustment Scale (WSAS) will be used to measure the daytime functioning of the participants such as ability to work, home management, social and private leisure activities, and close relationship maintenance.

CONTACTS AND LOCATIONS:
Overall Officials: Yun Kwok Wing, FRCPsych, Principal Investigator — Department of Psychiatry, the Chinese University of Hong Kong
Locations (1):
- Department of Psychiatry, the Chinese University of Hong Kong, Shatin, New Territories, Hong Kong

IPD SHARING:
Plan to Share IPD: No